CLINICAL TRIAL: NCT06497738
Title: A Prospective, Multi-center, Open-label, Cohort Study to Compare Daratumumab-Lenalidomide-Dexamethasone (DRd) With Modified Bortezomib-Lenalidomide-Dexamethasone (VRd-lite) in Elderly Newly Diagnosed Multiple Myeloma
Brief Title: A Prospective Study Comparing DRd With VRd-lite in Elderly Newly Diagnosed Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DRd
Record Dates: First submitted 2024-06-26; First posted 2024-07-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Daratumumab + lenalidomide + dexamethasone: Drug: Daratumumab Daratumumab will be administered at a dose of 16 milligram per kilogram (mg/kg) by intravenous (IV) infusion, once a week for 8 weeks, then once every other week for 16 weeks, thereafter once every 4 weeks. The total induction cycle is 8.
  Drug: Lenalidomide Lenalidomide will be self-administered at a dose of 25 mg orally on Day 1 to Day 21 of each 28-day cycle.
  Drug: Dexamethasone Dexamethasone 20 mg orally or intravenously on Days 1, 2, 8, 9, 15, 16, 22, 23 of each 21-day cycle for Cycles 1-8. For participant>75, dexamethasone will be reduced to 10mg twice a week.
  Then according to the risk stratification, standard risk participants will receive lenalidomide maintenance therapy while high risk participants will receive daratumumab combined with lenalidomide until progression.
- Modified Bortezomib+Lenalidomide+dexamethasone: Drug: Bortezomib Bortezomib 1.3 mg/m^2 will be administered by subcutaneous(SC) injection injection weekly on Days 1, 8, 15, 22 of each 21-day cycle for Cycles 1-8.
  Drug: Dexamethasone Dexamethasone 20 mg orally or intravenously on Days 1, 2, 8, 9, 15, 16, 22, 23 of each 21-day cycle for Cycles 1-8. For participant>75, dexamethasone will be reduced to 10mg twice a week.
  Then according to the risk stratification, standard risk participants will receive lenalidomide maintenance therapy while high risk participants will receive bortezomib combined with lenalidomide until progression.

SUMMARY:
The purpose of the study is to compare the efficacy and safety of daratumumab, lenalidomide and dexamethasone (DRd) to that of modified bortezomib, lenalidomide and dexamethasone (VRd-lite), in terms of progression-free survival and minimal residual disease negativity rate in elderly participants with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentered cohort study. This study will evaluate elderly participants with newly diagnosed multiple myeloma (MM) for whom hematopoietic stem cell transplant is not planned as initial therapy. All the eligible participants can be free to choose to receive either daratumumab lenalidomide and dexamethasone (DRd) or modified bortezomib lenalidomide and dexamethasone (VRd-lite). Daratumumab (16 milligram per kilogram [mg/kg]) will be administered weekly for first 8 weeks (Cycles 1 to 2) of treatment and then every other week for 16 weeks (Cycles 3 to 6), then every 4 weeks (Cycle 7 to 8). Bortezomib will be administered subcutaneously 1.3 mg/m^2 weekly of each 28-day cycle for Cycles 1-8. Lenalidomide will be administered at a dose of 25 mg orally on Days 1 through 21 of each 28-day cycle, and dexamethasone will be administered at a dose of 20 mg twice a week for both treatment arms. Participants in both treatment arms will continue at least lenalidomide maintenance until disease progression or unacceptable toxicity.The primary endpoint will be progression-free survival (PFS) and percentage of participants with Negative Minimal Residual Disease (MRD). Participant safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years old
2. Newly diagnosed Multiple myeloma patients with measurable disease. Diagnosis of multiple myeloma as documented per International Myeloma Working Group (IMWG) criteria：Monoclonal plasma cells in the bone marrow greater than or equal to (>=)10 percentage (%) or presence of a biopsy proven plasmacytoma and documented multiple myeloma satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or SLiM. CRAB criteria: Hypercalcemia: serum calcium greater than (>) 0.25 millimoles per liter (mmol/L) (>1 milligram per deciliter [mg/dL]) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL); Renal insufficiency: creatinine clearance less than (<) 40 milliliter per minute (mL/min) or serum creatinine >177 micro millimoles per liter (umol/L) (>2 mg/dL); Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL; Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography (PET)-CT. SLiM: Clonal bone marrow plasma cell percentage >=60%; Involved: uninvolved serum free light chain (FLC) ratio >=100; >1 focal lesion on magnetic resonance imaging (MRI) studies.

   Measurable disease: Immunoglobulin (Ig) G myeloma (serum monoclonal paraprotein [M-protein] level >= 0.5 gram/deciliter [g/dL] or urine M-protein level >= 200 milligram[mg]/24 hours[hrs]); OR IgA, IgM, IgD, or IgE multiple myeloma (serum M-protein level >= 0.2 g/dL or urine M-protein level >= 200 mg/24 hrs); OR Light chain multiple myeloma (serum immunoglobulin free light chain >= 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio)
3. Expected survival more than 3 months
4. No active infectious disease
5. Be able to understand the characteristics of the disease, voluntarily join this study protocol for treatment and follow-up
6. Have signed informed consent. Informed consent was obtained from the patients themselves or their immediate family members.

Exclusion Criteria:

1. Patients with active hepatitis B (HBV), hepatitis C (HCV), and other acquired, congenital immunodeficiency diseases.
2. Peripheral neuropathy or neuropathic pain(except extramedullary disease compression) Grade 2 or higher, as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.
3. Plasma cell leukemia, non-bone-related extramedullary lesions
4. Severe thrombotic events before treatment
5. The presence of grade 2 or higher peripheral neuropathy before treatment
6. Liver dysfunction (alanine aminotransferase and aspartate aminotransferase ≥ 2.5 times the upper limit of normal value)
7. Total bilirubin ≥ 1.5 times the upper limit of normal value
8. Major surgery within 30 days before enrollment
9. Epilepsy, dementia and other mental abnormalities requiring drug treatment and cannot understand or follow the study protocol
10. According to the protocol or the investigator's judgment, the patient has a serious physical or mental illness that may interfere with the participation in this clinical study
11. Drug abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or the evaluation of the study results
12. Patients who are receiving other experimental drug treatment
13. Lactating or pregnant women
14. The investigator believes that the participant is not suitable for enrollment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 1. Age ≥ 65 years old
  2. Newly diagnosed Multiple myeloma patients
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From enrollment to either disease progression or death whichever occurs first (approximately 5 years, or 8 years if the adaptive approach is decided at the interim)
  PFS is defined as the duration from date of enrollment to either progression disease(PD) or death, whichever comes first. International Myeloma Working Group (IMWG) criteria for PD: Increase of 25 percentage (%) from lowest response value in any one of following: Serum M-component (absolute increase must be >= 0.5 g/dL) Urine M-component (absolute increase must be >=200 mg/24 hours), participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain(FLC) levels (absolute increase must be >10 mg/dL), participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell(PC)% (absolute percentage must be >=10%), definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or tissue plasmacytomas and development of hypercalcemia (serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
MRD Negative Rate | First time reached VGPR, then12,18,24 Months and every 6 months
  Percentage of participants who have achieved MRD negative status will be assessed. MRD negativity will be evaluated as a potential surrogate for PFS and overall survival (OS) in multiple myeloma treatment.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Rate | Approximately 5 years
  VGPR or better rate is defined as the percentage of participants achieving VGPR and complete response (CR) (including stringent complete response [sCR]) prior to subsequent anti-myeloma therapy in accordance with the IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than or equal to (>=) 90 % reduction in serum M-protein plus urine M-protein <100 milligram per 24 hours (mg/24 hours); CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% PCs in bone marrow. sCR: CR plus normal FLC ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence or 2- to 4 color flow cytometry.
Overall Response Rate | Up to the end of the study (approximately 5 years)
  ORR is defined as the percentage of participants who achieve partial response (PR) or better responses prior to subsequent anti-myeloma therapy in accordance with IMWG criteria, during or after the study treatment. IMWG criteria for PR: greater than or equal to (>=) 50 reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90 % or to less than (<) 200 mg/24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow plasma cells (PCs) is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Duration of Response(DOR) | From initial documentation of response to the date of PD until approximately 5 years
  DOR is calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of PD, as defined in the IMWG evaluation before the start of any subsequent anti-myeloma therapy.
Overall Survival (OS) | From enrollment until the participant's death from any cause (up to approximately 5 years, or 8 years if the adaptive approach is decided at the interim)
  OS is defined as the time from the date of enrollment to the date of the participant's death due to any cause.
Complete Response (CR) or Better Rate | Approximately 5 years
  CR or better rate is defined as the percentage of participants achieving CR or sCR prior to subsequent anti-myeloma therapy in accordance with the IMWG criteria during or after the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Chen, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (6):
- China (6):
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu